CLINICAL TRIAL: NCT00505765
Title: A Multicenter Ascending Dose, Double Blind, Placebo-controlled Study of NAP (AL-108) in Chronic Schizophrenia
Brief Title: A Multicenter Study of NAP (AL-108) in Schizophrenia
Acronym: AL-108
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Maryland (Other); Washington University School of Medicine (Other); Massachusetts General Hospital (Other); Nathan Kline Institute for Psychiatric Research (Other); Columbia University (Other); Duke University (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TURNS03; HHSN 278200441003C (Other Grant/Funding Number: NIMH)
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Schizophrenia
Keywords: Cognition; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — davunetide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- AL-108, 30 mg/day (Experimental): AL-108, 30 mg/day- 3 sprays in each nostril, twice per day
  Interventions: Drug: AL-108
- AL-108, 5 mg/day (Experimental): AL-108, 5 mg/day- one spray in each nostril once per day
  Interventions: Drug: AL-108
- Placebo, 3 sprays BID (Placebo Comparator): Placebo- 3 sprays in each nostril, twice per day
  Interventions: Drug: Placebo
- Placebo, 1 Spray Daily (Placebo Comparator): Placebo- one spray in each nostril, once per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AL-108 — AL-108, 5 mg/day- one spray in each nostril once per day
  Arms: AL-108, 5 mg/day
Drug: AL-108 — AL-108, 30 mg/day- 3 sprays in each nostril, twice per day
  Arms: AL-108, 30 mg/day
Drug: Placebo — Placebo- 3 sprays in each nostril, twice per day
  Arms: Placebo, 3 sprays BID
Drug: Placebo — Placebo- one spray in each nostril, once per day
  Arms: Placebo, 1 Spray Daily

SUMMARY:
The TURNS is a NIMH-funded contract for the evaluation of new compounds for the treatment of cognitive impairments in schizophrenia (HHSN 27820044 1003C; P.I.: Steve Marder, M.D.). Despite advances in the safety, tolerability, and effectiveness of antipsychotic medications for the treatment of schizophrenia, many patients continue to be plagued by impairments in social and work functioning. Persons with schizophrenia commonly show deficits in a number of areas of cognition that include impairments in attention, memory, and executive functioning (the ability and organize one's behavior). Importantly, a large body of literature now shows a link between cognition and community functioning in schizophrenia. It is believed that treatments that improve cognitive deficits may lead to improvements in work and social functioning.

One approach to improve the community functioning of patients with schizophrenia is to develop new agents that treat the cognitive deficits of the illness. A promising agent is called AL-108. This drug is administered as a nasal spray. Studies in animals suggest that this drug may protect neurons and may improve cognition in schizophrenia. The current study is a twelve-week multicenter, double-blind, randomized clinical trial of two doses of AL-108 (5 and 30 mg/day intranasally) versus placebo in the treatment of persistent cognitive dysfunction in schizophrenia. The study medication will be added to patients' current atypical antipsychotic medication or to their current injectable first-generation antipsychotic medication. The primary outcome measure will consist of the composite score of the MATRICS neuropsychological battery. Secondary outcome measures will include scores on symptoms, functional outcome, and safety measures. Sixty clinically stable patients with schizophrenia, drawn from eight sites, will participate in the study. Twenty-five patients will be enrolled at UCLA.

DETAILED DESCRIPTION:
Background

AL-108 is an intranasal drug product containing NAP, an 8 amino-acid peptide (Asn-Ala-Pro-Val-Ser-Ile-Pro-Gln; NAPVSIPQ, MW=824.9) fragment of the much larger (approx. 124KD) Activity-Dependent Neuroprotective Protein (ADNP), which participates in neurodevelopment and neuroprotection. In mice, ADNP knockouts are lethal exhibiting CNS dysgenesis. ADNP mediates its effects in part through interaction with microtubules. Because of its large size, ADNP is assumed to not penetrate the BBB and thus cannot be used pharmacologically. NAP was chosen because it represents the epitope most associated with microtubule interaction and neuroprotection. NAP is absorbed following IV or intranasal administration, and has been shown to cross the BBB.

Rationale for NAP treatment: tubulin function in brain function

The cytoskeleton plays a key role in maintaining the highly asymmetrical shape and structural polarity of neurons that are essential for neuronal physiology. The cytoskeleton is made up of microfilaments, intermediate filaments and microtubules. Microfilaments (4-9 nm diameter) are made up of actin monomers and they function mainly to provide mechanical support and locomotion to the cell. Intermediate filaments are cytoplasmic fibers of ~10nm diameter. They provide supporting framework within the cell. Microtubules (~24nm diameter) consist of tubulin and microtubule associate proteins. They function to transport nutrients and chemical messengers along the cell. Neurofibrillary tangles are twisted bundles of neurofibrils formed when the microtubule-associated protein, tau, dissociates from microtubules and clusters to form an insoluble mass. Under normal conditions tau binds to microtubules, stabilizing neuronal structure and integrity.

Hyperphosphorylation of tau is assumed to be the cause for the formation of neurofibrillary tangles. Although neurofibrillary tangles are most associated with cognitive dysfunction in Alzheimers disease, some increase in neurofibrillary pathology has also been reported in schizophrenia, potentially as consequence of antipsychotic medication (1). Thus, mechanisms underlying microtubular function may be relevant to schizophrenia as well. In association with tubulin polymerization into microtubules, NAP influences tau dynamics by increasing the ratio of non-phosphorylated tau to phosphorylated tau, implying a dynamic process of cellular maintenance of the microtubular network, which is essential for the survival of the cell.

In brain, tubulin frameworks are stabilized by recently described STOP proteins (2) (aka MAP6). Linkages to allelic variation in STOP genes has been reported in schizophrenia, along with altered STOP protein expression in some brain regions (3). STOP knockdown mice show disturbances in dopaminergic neurotransmission (4) along with deficits in PPI and hypermotility that were partially reversed with clozapine (5). Thus, neuropathological features of schizophrenia may be due, in part, to abnormal STOP-related stabilization of microtubular structure, and NAP may stabilize STOP-related abnormal neurophysiological processes in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* DSM IV/DSM IV TR diagnosis of schizophrenia
* Capable of providing informed consent
* Males and Females
* Age: 18 and 60
* Caucasian or Non Caucasian
* Subjects will be treated with one of the following second generation antipsychotics: risperidone, olanzapine, quetiapine, ziprasidone, or aripiprazole for the previous two months, with no change in dose in the last month, and/or with injectable depot antipsychotics (fluphenazine or haloperidol decanoate) with no change in last 3 months.
* Subjects will meet the following symptom criteria:

  * Average Brief Psychiatric Rating Scale (BPRS) item score >3 (mild)
  * Simpson-Angus Scale total score less than or equal to 6
  * Calgary Depression Scale total score less than or equal to 10
* Subjects will meet the following cognitive performance criteria:

  * Performance less than the maximum cutoff (in parentheses) for ONE of the following MCCB tests:

    * Letter-number span (20);
    * HVLT total (31); and
    * CPT d-prime (3.47)
  * Able to complete the baseline MCCB validly as assessed by Chief Neuropsychologist or NP tester
  * Raw score of 6 or greater on the WTAR

Exclusion Criteria:

* Current treatment with oral conventional antipsychotics (e.g. fluphenazine, haloperidol) or clozapine.
* Subjects with a DSM-IV diagnosis of alcohol or substance abuse (other than nicotine) within the last month or a DSM-IV diagnosis of alcohol or substance dependence (other than nicotine) within the last 6 months
* Subjects with a history of significant head injury/trauma, as defined by one or more of the following:

  * Loss of consciousness (LOC) for more than 1 hour
  * Recurring seizures resulting from the head injury
  * Clear cognitive sequellae of the injury
  * Cognitive rehabilitation following the injury
* Subjects with a clinically significant neurological, metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, and/or urological disorder (e.g. unstable angina, decompensated congestive heart failure, CNS infection or history of HIV seropositivity), which would pose a risk to the patient if they were to participate in the study or that might confound the results of the study.
* Clinically significant abnormalities in physical examination, ECG, or laboratory assessments.
* Clinically significant renal disease.
* Women who are pregnant or of child-bearing potential, either not surgically-sterile nor using appropriate methods of birth control
* Women who are breast-feeding
* Prior participation in a clinical trial of investigational medication within 60 days.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2007-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Javitt, MD, PhD, Principal Investigator — Nathan Kline Institute
Locations (8):
- United States (8):
  - UCLA, Los Angeles, California
  - Maryland Psychiatric Research Center, Catonsville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Harvard Medical School, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Nathan Kline Institute, Orangeburg, New York
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Background] McMahon RP, Arndt S, Conley RR. More powerful two-sample tests for differences in repeated measures of adverse effects in psychiatric trials when only some patients may be at risk. Stat Med. 2005 Jan 15;24(1):11-21. doi: 10.1002/sim.1837. PMID 15515151
- [Background] Edwards D, Madsen J. Constructing multiple test procedures for partially ordered hypothesis sets. Stat Med. 2007 Dec 10;26(28):5116-24. doi: 10.1002/sim.2905. PMID 17476650
- [Background] Jackman AH, Doty RL. Utility of a three-item smell identification test in detecting olfactory dysfunction. Laryngoscope. 2005 Dec;115(12):2209-12. doi: 10.1097/01.mlg.0000183194.17484.bb. PMID 16369168
- [Background] Gozes I, Divinski I. The femtomolar-acting NAP interacts with microtubules: Novel aspects of astrocyte protection. J Alzheimers Dis. 2004 Dec;6(6 Suppl):S37-41. doi: 10.3233/jad-2004-6s605. PMID 15665412
- [Background] Rothermundt M, Arolt V, Bayer TA. Review of immunological and immunopathological findings in schizophrenia. Brain Behav Immun. 2001 Dec;15(4):319-39. doi: 10.1006/brbi.2001.0648. PMID 11782102
- [Background] Rapaport MH, Delrahim KK. An abbreviated review of immune abnormalities in schizophrenia. CNS Spectr. 2001 May;6(5):392-7. doi: 10.1017/s1092852900021763. PMID 15999027
- [Background] Kelly DL, Conley RR. A randomized double-blind 12-week study of quetiapine, risperidone or fluphenazine on sexual functioning in people with schizophrenia. Psychoneuroendocrinology. 2006 Apr;31(3):340-6. doi: 10.1016/j.psyneuen.2005.08.010. Epub 2005 Sep 28. PMID 16198059
- [Background] Gozes I, Meltzer E, Rubinrout S, Brenneman DE, Fridkin M. Vasoactive intestinal peptide potentiates sexual behavior: inhibition by novel antagonist. Endocrinology. 1989 Dec;125(6):2945-9. doi: 10.1210/endo-125-6-2945. PMID 2583049
- [Background] Rotstein M, Bassan H, Kariv N, Speiser Z, Harel S, Gozes I. NAP enhances neurodevelopment of newborn apolipoprotein E-deficient mice subjected to hypoxia. J Pharmacol Exp Ther. 2006 Oct;319(1):332-9. doi: 10.1124/jpet.106.106898. Epub 2006 Jul 5. PMID 16822898
- [Background] Oddo S, Caccamo A, Shepherd JD, Murphy MP, Golde TE, Kayed R, Metherate R, Mattson MP, Akbari Y, LaFerla FM. Triple-transgenic model of Alzheimer's disease with plaques and tangles: intracellular Abeta and synaptic dysfunction. Neuron. 2003 Jul 31;39(3):409-21. doi: 10.1016/s0896-6273(03)00434-3. PMID 12895417
- [Background] Braga RJ, Mendlowicz MV, Marrocos RP, Figueira IL. Anxiety disorders in outpatients with schizophrenia: prevalence and impact on the subjective quality of life. J Psychiatr Res. 2005 Jul;39(4):409-14. doi: 10.1016/j.jpsychires.2004.09.003. Epub 2004 Nov 13. PMID 15804391
- [Background] Alcalay RN, Giladi E, Pick CG, Gozes I. Intranasal administration of NAP, a neuroprotective peptide, decreases anxiety-like behavior in aging mice in the elevated plus maze. Neurosci Lett. 2004 May 6;361(1-3):128-31. doi: 10.1016/j.neulet.2003.12.005. PMID 15135910
- [Background] Gozes I, Alcalay R, Giladi E, Pinhasov A, Furman S, Brenneman DE. NAP accelerates the performance of normal rats in the water maze. J Mol Neurosci. 2002 Aug-Oct;19(1-2):167-70. doi: 10.1007/s12031-002-0028-0. PMID 12212775
- [Background] Gozes I, Giladi E, Pinhasov A, Bardea A, Brenneman DE. Activity-dependent neurotrophic factor: intranasal administration of femtomolar-acting peptides improve performance in a water maze. J Pharmacol Exp Ther. 2000 Jun;293(3):1091-8. PMID 10869414
- [Background] Ito M, Depaz I, Wilce P, Suzuki T, Niwa S, Matsumoto I. Expression of human neuronal protein 22, a novel cytoskeleton-associated protein, was decreased in the anterior cingulate cortex of schizophrenia. Neurosci Lett. 2005 Apr 22;378(3):125-30. doi: 10.1016/j.neulet.2004.12.079. PMID 15781144
- [Background] Benitez-King G, Ramirez-Rodriguez G, Ortiz L, Meza I. The neuronal cytoskeleton as a potential therapeutical target in neurodegenerative diseases and schizophrenia. Curr Drug Targets CNS Neurol Disord. 2004 Dec;3(6):515-33. doi: 10.2174/1568007043336761. PMID 15581421
- [Background] Kolluri N, Sun Z, Sampson AR, Lewis DA. Lamina-specific reductions in dendritic spine density in the prefrontal cortex of subjects with schizophrenia. Am J Psychiatry. 2005 Jun;162(6):1200-2. doi: 10.1176/appi.ajp.162.6.1200. PMID 15930070
- [Background] Hill JJ, Hashimoto T, Lewis DA. Molecular mechanisms contributing to dendritic spine alterations in the prefrontal cortex of subjects with schizophrenia. Mol Psychiatry. 2006 Jun;11(6):557-66. doi: 10.1038/sj.mp.4001792. PMID 16402129
- [Background] Harrison PJ. The neuropathology of schizophrenia. A critical review of the data and their interpretation. Brain. 1999 Apr;122 ( Pt 4):593-624. doi: 10.1093/brain/122.4.593. PMID 10219775
- [Background] Smith-Swintosky VL, Gozes I, Brenneman DE, D'Andrea MR, Plata-Salaman CR. Activity-dependent neurotrophic factor-9 and NAP promote neurite outgrowth in rat hippocampal and cortical cultures. J Mol Neurosci. 2005;25(3):225-38. doi: 10.1385/JMN:25:3:225. PMID 15800376
- [Background] Fradley RL, O'Meara GF, Newman RJ, Andrieux A, Job D, Reynolds DS. STOP knockout and NMDA NR1 hypomorphic mice exhibit deficits in sensorimotor gating. Behav Brain Res. 2005 Sep 8;163(2):257-64. doi: 10.1016/j.bbr.2005.05.012. PMID 16046005
- [Background] Brun P, Begou M, Andrieux A, Mouly-Badina L, Clerget M, Schweitzer A, Scarna H, Renaud B, Job D, Suaud-Chagny MF. Dopaminergic transmission in STOP null mice. J Neurochem. 2005 Jul;94(1):63-73. doi: 10.1111/j.1471-4159.2005.03166.x. PMID 15953350
- [Background] Shimizu H, Iwayama Y, Yamada K, Toyota T, Minabe Y, Nakamura K, Nakajima M, Hattori E, Mori N, Osumi N, Yoshikawa T. Genetic and expression analyses of the STOP (MAP6) gene in schizophrenia. Schizophr Res. 2006 Jun;84(2-3):244-52. doi: 10.1016/j.schres.2006.03.017. Epub 2006 Apr 19. PMID 16624526
- [Background] Bosc C, Andrieux A, Job D. STOP proteins. Biochemistry. 2003 Oct 28;42(42):12125-32. doi: 10.1021/bi0352163. PMID 14567673
- [Background] Harrison PJ. The neuropathological effects of antipsychotic drugs. Schizophr Res. 1999 Nov 30;40(2):87-99. doi: 10.1016/s0920-9964(99)00065-1. PMID 10593448
- [Derived] Georgiades A, Davis VG, Atkins AS, Khan A, Walker TW, Loebel A, Haig G, Hilt DC, Dunayevich E, Umbricht D, Sand M, Keefe RSE. Psychometric characteristics of the MATRICS Consensus Cognitive Battery in a large pooled cohort of stable schizophrenia patients. Schizophr Res. 2017 Dec;190:172-179. doi: 10.1016/j.schres.2017.03.040. Epub 2017 Apr 20. PMID 28433500

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 of 69 randomized participants were excluded prior to starting medication
Groups:
- Placebo: Placebo, low-dose: 1 puff administered in each nostril daily (QD) Placebo, high-dose: 3 puffs administered twice daily in each nostril (BID)
  Data were combined across placebo conditions for analysis
Period: Overall Study
Arm/Group | AL-108, 30 mg/Day | AL-108, 5 mg/Day | Placebo
Started | 21 | 20 | 22
Mid-Point Assessment | 20 | 19 | 21
Completed | 19 | 17 | 19
Not Completed | 2 | 3 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Noncompliance | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Of 69 randomized participants, 6 were excluded prior to starting double-blind medication; 63 participants exposed to drug or placebo were included in analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | AL-108, 30 mg/Day | AL-108, 5 mg/Day | Placebo | Total
Number analyzed (Participants) | 21 | 20 | 22 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (8.2) | 43.2 (10.5) | 41.4 (10.4) | 43.4 (10.2)
Sex/Gender, Customized [Number; unit: participants]
  Female | 7 | 7 | 8 | 22
  Male | 14 | 13 | 14 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 8 | 22
  Male | 14 | 13 | 14 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity
  Participants
    Hispanic | 0 | 3 | 1 | 4
    Non-Hispanic | 21 | 17 | 21 | 59

OUTCOME MEASURES:

1. Primary Outcome: Change in MATRICS Consensus Cognitive Battery Composite Score Change
Description: The MATRICS Consensus Cognitive Battery (MCCB) measures functioning across various cognitive domains and is comprised of ten tests that assess seven cognitive domains (speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition) Its measurements are based on timed paper-and-pencil, computerized, and orally-administered tests, as well as spatial tests using geometric cubes. MCCB composite T scores are between 40 and 60 (normal range) and < 40 (below normal range).
Time Frame: Baseline, week 6
Population: Only participants with completed MCCB at both baseline and 6 weeks were included in analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AL-108, 30 mg/Day | AL-108, 5 mg/Day | Placebo
Number analyzed (Participants) | 19 | 19 | 20
units on a scale | 1.3 (4.6) | 2.3 (4.6) | -0.2 (5.6)

2. Primary Outcome: Change in MATRICS Consensus Cognitive Battery (MCCB)
Description: as for outcome 1
Time Frame: Baseline, 12 weeks
Population: Only participants with completed MCCB at both Baseline and 12 weeks were included in analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AL-108, 30 mg/Day | AL-108, 5 mg/Day | Placebo
Number analyzed (Participants) | 18 | 17 | 19
units on a scale | 3.9 (4.6) | 4.6 (7.2) | 3.2 (4.9)
Statistical Analysis 1: Comparison: AL-108, 5 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.21, ANCOVA; Mean Difference (Final Values) = 1.9, Standard Deviation 1.5
Statistical Analysis 2: Comparison: AL-108, 30 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.44, ANCOVA; Mean Difference (Final Values) = 1.2, Standard Deviation 1.5

3. Secondary Outcome: Change in UCSD Performance-Based Skills Assessment (UPSA) Summary Scores
Description: UPSA includes 5 skill areas (subscales) with scores that each range from 0-20. The UPSA yields an overall total score which is the sum of the five subscales and ranges from 0-100. Higher scores are associated with more independent living.
Time Frame: Baseline, week 6
Population: Only participants with UPSA scores at both Baseline and 6 weeks were included in this analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AL-108, 30 mg/Day | AL-108, 5 mg/Day | Placebo
Number analyzed (Participants) | 20 | 19 | 19
units on a scale | 2.9 (7.6) | 7.2 (7.3) | -0.9 (9.0)

4. Secondary Outcome: Change in UCSD Performance-Based Skills Assessment (UPSA) Summary Scores
Description: as for outcome 3
Time Frame: Baseline, 12 weeks
Population: Only participants with UPSA scores at both Baseline and 12 weeks were included in this analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AL-108, 30 mg/Day | AL-108, 5 mg/Day | Placebo
Number analyzed (Participants) | 19 | 17 | 18
units on a scale | 4.9 (19) | 8.9 (6.6) | 0.3 (8.5)

5. Secondary Outcome: Change in SCoRS Interviewer Global Rating
Description: Schizophrenia Cognition Rating Scale (SCoRS) assessed functional capacity by completing a 20-question rating scale via interviews with the subject and an informant, focusing on cognitive impairment and its impact on daily functioning. After the interview, the interviewer rated subject's overall difficulty on a Global Scale of 1-10. Higher scores indicate greater cognitive impairment.
Time Frame: Baseline, 6 weeks
Population: Participants administered SCoRS at both Baseline and 6 weeks were included in analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AL-108, 30 mg/Day | AL-108, 5 mg/Day | Placebo
Number analyzed (Participants) | 16 | 17 | 21
units on a scale | 0.1 (1.2) | -0.6 (1.3) | -0.1 (1.0)

6. Secondary Outcome: Change in SCoRS Interviewer Global Rating
Description: as for outcome 5
Time Frame: Baseline, 12 weeks
Population: Participants administered SCoRS at both Baseline and 12 weeks were included in analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AL-108, 30 mg/Day | AL-108, 5 mg/Day | Placebo
Number analyzed (Participants) | 16 | 16 | 18
units on a scale | -0.4 (1.1) | -1.2 (1.6) | -0.3 (1.5)

ADVERSE EVENTS:
Description: Of 69 randomized participants, 6 were excluded prior to starting double-blind medication; 63 participants exposed to drug or placebo were included in analyses.
Arm/Group | AL-108, 30 mg/Day | AL-108, 5 mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/20 | 0/22
Other Adverse Events (participants affected / at risk) | 4/21 | 9/20 | 2/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AL-108, 30 mg/Day (N=21) | AL-108, 5 mg/Day (N=20) | Placebo (N=22)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Pt was hospitalized overnight for palpitations.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AL-108, 30 mg/Day (N=21) | AL-108, 5 mg/Day (N=20) | Placebo (N=22)
Restlessness (Nervous system disorders) | 4 (4) | 9 (9) | 2 (2) — Self-reported restlessness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No